CLINICAL TRIAL: NCT02055404
Title: On-Eye Evaluation of Contact Lens Rotation Marks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: C-12-045
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-02

CONDITIONS: Refractive Error
Keywords: astigmatism; toric; contact lenses; daily disposable contact lenses; molded mark; rotation mark
MeSH Terms: conditions — Refractive Errors; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delefilcon A (Experimental): Delefilcon A spherical contact lens with molded marks randomly assigned to one eye, with etafilcon A toric contact lens in the fellow eye for contralateral wear approximately 2 hours in duration
  Interventions: Device: Delefilcon A spherical contact lens with molded marks
- Etafilcon A (Other): Etafilcon A toric contact lens randomly assigned to one eye, with delefilcon A spherical contact lens with molded marks in the fellow eye for contralateral wear approximately 2 hours in duration
  Interventions: Device: Etafilcon A toric contact lens

INTERVENTIONS:
Device: Delefilcon A spherical contact lens with molded marks — Silicone hydrogel contact lens with 9 different molded marks of varying widths and depths indented into the front surface (S1, S2, S3, S4, S5, S6, S7, S8, and S9). Each lens contained all 9 marks.
  Arms: Delefilcon A
Device: Etafilcon A toric contact lens — Hydrogel toric contact lens for daily wear, daily disposable use
  Other Names: 1-DAY ACUVUE® MOIST® for ASTIGMATISM
  Arms: Etafilcon A

SUMMARY:
The purpose of this study was to select the size of the molded rotation mark for a new toric contact lens by comparing the visibility of various molded rotation marks.

DETAILED DESCRIPTION:
Participants wore the test and control products contralaterally (in each eye separately) for 2 hours, during which the Investigator assessed the various molded rotation marks for visibility. Each participant was assessed by 10 investigators.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent document.
* Best corrected distance visual acuity (VA) greater than or equal to 20/25 in each eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* History of any ocular surgery or ocular injury within 12 weeks of study enrollment.
* Any ocular disease, infection, inflammation, or abnormality that contraindicates contact lens (CL) wear.
* History of herpetic keratitis.
* Slit-lamp findings greater than grade 2 at baseline.
* Any use of systemic or ocular medications for which CL wear could be contraindicated.
* Inactive corneal neovascularization greater than 1 millimeter of penetration.
* A clinically significant dry eye not responding to treatment.
* History of refractive surgery.
* Participation in a clinical study within the previous 30 days.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Nick, Dipl. Ing., Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 US study center.
Pre-assignment Details: This reporting group includes all enrolled participants.
Groups:
- Overall Study: Delefilcon A spherical contact lens with molded marks and etafilcon A toric contact lens worn contralaterally (1 in each eye) for approximately 2 hours
Period: Overall Study
Arm/Group | Overall Study
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The analysis population includes all enrolled participants.
Arm/Group | Overall Study
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (21.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Visibility of Rotation Mark (Clearly Visible, Slightly Visible Acceptable)
Description: Each lens (containing 8 rotation marks and one reference mark, in total 9 marks) was assessed for visibility by 10 investigators using the following scale: "N/A;" "Not visible;" "Slightly visible, not acceptable;" "Slightly visible, acceptable;" "Clearly visible;" "More visible than necessary." Visibility assessments were made after all marks had been evaluated. S9 Mark (test lens) functioned as a starting marker only and was not rated. The control lens was not used as a comparison, but rather as a reference for what a mark looks like on a commercial product. "Visibility of Rotation Mark" is reported as the percentage of assessments rating the rotation mark as "Clearly visible" or "Slightly visible, acceptable."
Time Frame: Day 1
Population: The analysis population includes all enrolled participants. Assessments from all 10 investigators were analyzed, hence sample size for each rotational mark is 30.
Measure: Number; unit: Percentage of assessments
Groups:
- S1 Mark; S2 Mark; S3 Mark; S4 Mark; S5 Mark; S6 Mark; S7 Mark; S8 Mark: Delefilcon A spherical contact lens with 1 of 9 molded marks
- Control: Etafilcon A toric contact lens
Arm/Group | S1 Mark | S2 Mark | S3 Mark | S4 Mark | S5 Mark | S6 Mark | S7 Mark | S8 Mark | Control
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Percentage of assessments | 42.9 | 71.4 | 78.6 | 46.4 | 71.4 | 82.1 | 78.6 | 75.0 | 93.3

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (1 day).
Description: The analysis population includes includes all enrolled participants.
Arm/Group | Delefilcon A | Etafilcon A
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes